CLINICAL TRIAL: NCT05616949
Title: Peer Recovery Support Services for Individuals in Recovery Residences on MOUD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Potomac Health Foundations (Other)
Collaborators: National Institute of Drug Abuse (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA057627-01 (NIH)
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Opioid Use Disorder; Substance Use Disorder
Keywords: Medications for Opioid Use Disorder; Opioid Use Disorder; Recovery Residence; Peer Support; Intervention
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A parallel group randomized design is used. Participants will be randomized to receive treatment as usual (TAU) or the Peer Recovery Support Services (PRSS) intervention with a focus on MOUD retention. Individuals in the PRSS intervention group will receive all components of TAU plus additional peer-delivered recovery support services to aimed at enhancing retention in MOUD treatment. The plan is to recruit 50 total individuals. If there is significant drop out. Randomization will occur in a 1:1 ratio by flipping a coin, and will be conducted using stratified block randomization using random block sizes. Gender is the only stratification variable. Study staff involved with recruitment will be blinded to the participant's condition until after randomization. After randomization, the participant and study staff will all know if the participant was randomized to TAU or to PRSS. The intervention period is 24-weeks with follow ups at weeks 36 and 52.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 Title: Treatment as Usual (TAU) (Active Comparator): Arm 1: Treatment as Usual (TAU): The treatment and/or other services received as part of usual care while living in a recovery residence. This arm serves as the active comparator group for the study.
  Interventions: Behavioral: Treatment as Usual (TAU) (Arm 1)
- Arm 2 Title: Peer Recovery Support Services (PRSS) + TAU (Experimental): Arm 2: Peer Recovery Support Services (PRSS) Intervention: The experimental group for this study that involves the implementation of the PRSS intervention. This study will test the preliminary efficacy of the PRSS intervention on Medications for Opioid Use Disorder (MOUD) retention by evenly randomizing N=50 individuals on MOUD living in recovery residences (RRs) to either a 24-week course of the experimental PRSS intervention layered on top of treatment as usual services (TAU+PRSS) vs. an active comparator composed of treatment as usual services without the PRSS intervention (i.e., TAU-alone). Follow ups will be conducted at weeks 2, 4, 8, 12, 16, 20, 24 (end of intervention), 36, and 52 to collect data on the primary outcome of MOUD retention and other outcomes.
  Interventions: Behavioral: Peer Recovery Support Services (PRSS) + TAU (experimental- Arm 2)

INTERVENTIONS:
Behavioral: Treatment as Usual (TAU) (Arm 1) — Treatment as Usual (TAU): The treatment and/or other services received as part of usual care while living in a recovery residence. This arm serves as the active comparator group for the study.
  Arms: Arm 1 Title: Treatment as Usual (TAU)
Behavioral: Peer Recovery Support Services (PRSS) + TAU (experimental- Arm 2) — Peer Recovery Support Services (PRSS) Intervention: The experimental group for this study that involves the implementation of the PRSS intervention. This study will test the preliminary efficacy of the PRSS intervention on Medications for Opioid Use Disorder (MOUD) retention by evenly randomizing N=50 individuals on MOUD living in recovery residences (RRs) to either a 24-week course of the experimental PRSS intervention layered on top of treatment as usual services
  Arms: Arm 2 Title: Peer Recovery Support Services (PRSS) + TAU

SUMMARY:
The United States is experiencing an unprecedented opioid epidemic with a rapid increase in overdose deaths. Medications for opioid use disorder (MOUD) including methadone, buprenorphine, and extended-release naltrexone are efficacious and the recommended standard of care, yet barriers to sustained MOUD treatment reduce the overall efficacy of MOUD. Rates of MOUD retention are alarmingly low and MOUD dropout predicts opioid use/relapse, overdose, and death. While previous research has identified predictors of MOUD retention and adherence, there are no evidence-based interventions to improve MOUD retention.

Recovery support services are a broad set of strategies to promote healthy outcomes among individuals with substance use disorder (SUD) that are typically separate from standard professional treatment. Among those strategies most utilized are peer recovery support services (PRSS) and recovery residences (RRs). PRSS include coaching, mentoring, education, and other supports delivered by individuals uniquely qualified by their lived experience with SUD. PRSS are increasingly utilized in a range of clinical settings, and advantages of PRSS include inherent shared understanding of addiction and a high degree of acceptance and understanding that is not found in most professional relationships. Existing research tentatively supports PRSS; however, the evidence to date is sparse and comes with significant methodological limitations and inconsistencies that make it difficult to conclude the efficacy of PRSS. No studies have examined the role of PRSS in promoting retention in MOUD. RRs provide a supportive living environment for persons in recovery from SUD and are widely utilized in the United States with an estimated 17,943 residences in 2020. Despite their proliferation, the evidence for RRs is only moderate and diminished by methodological weaknesses. Further, individuals on MOUD seeking housing through RRs often face increased MOUD-related stigma or may be disqualified from a RR for taking MOUD and need additional support to navigate these challenges.

The potential synergistic benefits of combining PRSS and RRs to improve MOUD retention are considerable. PRSS and RRs are already mainstays in the recovery support services repertoire and could be leveraged to support MOUD retention. For example, more frequent, informal outreach typical of PRSS could facilitate regular monitoring of shifting attitudes and behaviors related to MOUD. The structure and accountability embedded in RRs could be used to support MOUD adherence and retention. Waxing and waning motivation to participate in MOUD treatment is common, and standard treatment is often unsuccessful at identifying early signs of future dropout or facilitating re-engagement after dropout.

We will recruit participants on MOUD in RRs and provide them with PRSS using approaches such as recovery coaching and care navigation with a particular focus on supporting retention in MOUD care. PRSS will also provide assertive outreach between episodes of care, emphasize continuation in treatment and other recovery activities after leaving a RR (either successfully or unsuccessfully), and emphasize return to care after treatment dropout and/or relapse. The peers will be deeply embedded within the local provider community and care continuum to facilitate ease of care navigation. The ultimate goal of our research agenda is to test the efficacy of a PRSS intervention among individuals with OUD living in RRs through a rigorous trial. The eventual trial design would be informed by preparatory activities and experience proposed in this planning project.

Preparatory activities proposed in this project include three major phases. Phase 1 - preparation for the intervention including: building a network of RRs that will be recruitment sites in the pilot RCT, recruiting and training peer support specialists, conducting focus groups and interviews to gather stakeholder input, and developing PRSS approaches to promote MOUD retention. Phase 2 - pilot test the PRSS intervention by randomizing N=50 individuals on MOUD recruited from collaborating RRs to either: a 24-week course of the PRSS intervention added to usual services, or usual services without the PRSS intervention. Phase 3 - gather additional input from former participants and RR staff post-intervention to further refine the intervention, and use lessons learned to inform our trial design and data collection procedures for the next-step R01 application.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ (inclusive); meets diagnostic criteria for OUD; residing at a RR affiliated with this study; seeking treatment with and successfully inducted onto MOUD (i.e., XR-NTX, SL-BUP, XR-BUP, or methadone); English speaking; willing and able to provide informed consent.

Exclusion Criteria:

* Currently receiving formalized PRSS outside of the study (not applicable to peer support typical of sponsorship in 12-step mutual support programs or informal support through RRs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
cumulative MOUD retention | Cumulative MOUD Retention is the proportion of days on MOUD at 24-weeks (end of intervention period).
  Primary Outcome: Cumulative MOUD retention on all follow-up assessments for the following data sources: 1) Time Line Follow Back; 2) the Maryland PDMP; and 3) Patient Health Records.

SECONDARY OUTCOMES:
Secondary Outcome 1- continuous MOUD retention ("yes" or "no") | Participants who are continuously retained have no gaps in MOUD exceeding 14-days.
  Continuous MOUD retention on all follow-up assessments will be tracked for the following data sources: 1) Time Line Follow Back; 2) the Maryland PDMP; and 3) Patient Health Records.
Secondary Outcome 2- opioid relapse ("yes" or "no") | Relapse is defined as ten days of use within a 4-week period.
  Opioid relapse are measured by tracking responses on the following data sources: Time Line Follow Back.
Secondary Outcome 3- re-initiation of MOUD after dropout ("yes" or "no") | Re-initiation of MOUD is defined as re-initiation onto any MOUD for at least 7 days after MOUD dropout (defined as >14 days without MOUD).
  Re-initiation of MOUD after dropout will be measured by examining all follow-up assessments after dropout for the following data sources: 1) Time Line Follow Back; 2) the Maryland PDMP; and 3) Patient Health Records.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R. Wenzel, Ph.D., Principal Investigator — Mountain Manor Treatment Center - Maryland Treatment Centers; Marc J. Fishman, M.D., Principal Investigator — Mountain Manor Treatment Center - Maryland Treatment Centers
Locations (2):
- United States (2):
  - Maryland Treatment Centers, Baltimore, Maryland
  - Maryland Treatment Centers/Avery Road Treatment Center, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: No